CLINICAL TRIAL: NCT02811718
Title: Resiliency Training for Patients With Neurofibromatosis Via Videoconferencing With Skype
Brief Title: Resiliency Training for Patients With NF2 Via Videoconferencing With Skype
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: The Children's Tumor Foundation (Other)
Responsible Party: Principal Investigator, Ana-Maria Vranceanu, PhD, Clinical Psychologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013P002605b
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Neurofibromatosis 2
Keywords: Stress Management; Resiliency; Skype
MeSH Terms: conditions — Neurofibromatosis 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stress Management Group 1 (Experimental): Subjects will attend group stress management sessions via Skype once weekly for 8 weeks and learn stress/NF symptoms managements techniques.
  Interventions: Behavioral: Stress Management Group 1
- Stress Management Group 2 (Experimental): Subjects will attend group stress management sessions via Skype once weekly for 8 weeks and learn stress/NF symptoms managements techniques.
  Interventions: Behavioral: Stress Management Group 2

INTERVENTIONS:
Behavioral: Stress Management Group 1 — Subjects will attend group stress management sessions via Skype once weekly for 8 weeks and learn stress/NF symptoms managements techniques.
  Arms: Stress Management Group 1
Behavioral: Stress Management Group 2 — Subjects will attend group stress management sessions via Skype once weekly for 8 weeks and learn stress/NF symptoms managements techniques.
  Arms: Stress Management Group 2

SUMMARY:
The aim of this study is to determine, whether the 3RP is feasible, accepted and efficacious and durable when delivered via Skype to patients with neurofibromatosis type 2 (NF2) who are deaf or have severe hearing loss using Communication Access Realtime Translation (CART) and/or American Sign Language (ASL).

This will be a substudy of the IRB-approved protocol #2013P002605. It is the same study except it is looking at a particular sub-population: patients with NF2 who are hard of hearing.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Can read and speak English at or above the 6th grade level
3. Patients with NF2 who are deaf or have severe hearing loss.

Exclusion Criteria:

1. Severe active or untreated major mental illness that would interfere with study participation, to be determined at the discretion of the study investigator (e.g. untreated psychosis or suicidality)
2. Recent (within past 3 months) change in antidepressant medication
3. Use of formal relaxation training (including past participation in a mind-body program), currently or in the past 6 months.
4. Unable or unwilling to sign the informed consent documents
5. Unable or unwilling to complete psychological assessments online via the REDCap system.
6. Unable or unwilling to participate in an intervention delivered via videoconferencing with Skype.
7. Unwilling to use either CART or ASL for communication during the Skype groups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Quality of Life (WHOQOL-BREF) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32 and week 64)
  The WHOQOL-BREF comprises of 26 items which measure the following broad domains: physical health, psychological health, social relationships, and environment. The WHOQOL-BREF is a shorter version of the original instrument that may be more convenient for use in large research studies or clinical trials.
Penn Acoustic Neuroma Quality-of Life Scale (PANQOL) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32 and week 64)
  The PANQOL measures quality of life specifically for patients with NF2.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS-10) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The PSS is a widely used psychological instrument for the measurement of the perception of stress. This 10-itam scale is designed to measure the degree to which situations in one's life are appraised, or considered stressful. The scores range from 0-40, with a higher score indicating higher perceived stress. Items were designed to detect how unpredictable, uncontrollable and overloaded respondents find their lives.
The 14-Item Resiliency Scale (RS-14) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The RS-14 measures stress coping ability in the face of adversity.
Patient Health Questionnaire (PHQ) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The PHQ measures symptoms of depression and functional impairment.
Cognitive and Affective Mindfulness Scale (CAMS) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The CAMS measures the degree to which individuals experience their thoughts and feelings.
Life Orientation Test (LOT) Optimism Scale | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The LOT Optimism Scale measures individual differences in generalized optimism versus pessimism.
The Gratitude Questionnaire (GQ-6) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The GQ-6 revised is a 6-item measure that assesses individual differences in the proneness to experience gratitude in daily life. Scores range from 6-42, with a higher score indicating a greater sense of gratitude.
Measure of Current Status (MOCS-A) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The MOCS-A is a 13-item measure assessing participants' current self-perceived status on several skills such as: the ability to relax at will, recognize stress-inducing situations, restructure maladaptive thoughts, be assertive about needs, and choose appropriate coping responses as needed. Responses are made on a 7-point scale with higher scores reflecting higher life satisfaction.
Medical Outcomes Study (MOS) Social Support Survey | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The MOS Social Support Survey measures various dimensions of social support.

OTHER OUTCOMES:
Intent to Attend | Baseline (week 0)
  Measures how likely and how motivated the participants is to attend the next session.
Date of Birth, Age, Gender, Race, Ethnicity, Marital Status, Education Status, Employment Status, and hearing status of subjects with NF2 | Baseline (week 0)
  This questionnaire asks subjects with NF2 to report their date of birth, age, gender, race, ethnicity, marital status, highest level of education, hearing status, and primary employment status over the last 12 months.
Credibility Questionnaire | Baseline (week 0)
  Measures how much the participant believes the intervention will work.
Client Satisfaction Questionnaire (CSQ-8) | Post-intervention (week 8)
  Measures how satisfied the participant is with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Maria Vranceanu, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided